CLINICAL TRIAL: NCT06620380
Title: Ex Vivo Drug Response Evaluation for Next Generation Care of Brain Metastases
Acronym: EViDENCE-BM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: anticancerfund.org (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EViDENCE-BM
Record Dates: First submitted 2024-05-27; First posted 2024-10-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastases; Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase II interventional randomized non-comparative clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (2):
- Arm 1: experimental arm, Pharmacoscopy-guided treatment (Experimental): Arm 1 (experimental arm): Pharmacoscopy-guided treatment will be prescribed by the investigator according to the results of the analysis (relevant on-target effect) and per drug prescription guidelines.
  Interventions: Device: Pharmacoscopy 1.0
- Arm 2: control arm (Active Comparator): For patients randomized to the control arm, no pharmacoscopy analysis will be performed.
  Interventions: Other: Control

INTERVENTIONS:
Device: Pharmacoscopy 1.0 — Pharmacoscopy is currently an academically developed platform. The study is designed to investigate the clinical performance of this academic platform. In the interventional arm, the best candidate agent defined by pharmascopy will be considered to guide the therapeutic decision for each patient.
  Arms: Arm 1: experimental arm, Pharmacoscopy-guided treatment
Other: Control — The next systemic treatment after surgery will be discussed, with the investigator and at the tumor board, considering also standard histopathological and molecular analysis, including next generation sequencing, molecular profiling analysis and previous treatments received
  Arms: Arm 2: control arm

SUMMARY:
Pharmacoscopy refers to an ex vivo real-time drug sensitivity profiling platform that has been shown to be of value in the treatment of leukemia (Snijder et al. 2017) (Kornauth et al. 2022) and may help to identify novel treatment opportunities for brain tumors as well (Lee et al. 2022). The rationale for pharmacoscopy-based drug sensitivity testing on real-time patient biopsies or surgery material is multiple: measuring drug response and sensitivity directly in real-time patient material, overcomes the problem of limited molecular biomarkers for established targeted therapeutic options and can identify effective drugs even for non-targeted therapies such as chemotherapy. It can also identify hitherto unknown specific vulnerabilities of cancer cells. Furthermore, testing directly on patient material overcomes the limitations of patient-derived cell cultures, organoids, and patient xenografts, as their prolonged culture times risk cellular adaptations and clonal selection that alter drug sensitivity. Pharmacoscopy maintains the tumor cell composition, including bystander cells or tumor microenvironment, and limits cell culture to max 48 hours. Furthermore, pharmacoscopy measures drug responses on a single-cell and on a high-content level, uniquely allowing to measure the drug sensitivity of tumor cells, and allowing to compare it to the drug cytotoxicity on healthy cells from the same patient. This relative readout has previously been shown to be essential for the correct prediction of a clinical response in haematological malignancies (Snijder et al. 2017) (Kornauth et al. 2022).

The aim of this study is to generate preliminary data regarding superiority of the personalized pharmacoscopy-guided approach compared to a standard non-pharmacoscopy-guided approach, in patients with brain metastases with an indication for surgery, and limited therapeutic systemic options according to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older on the day of signing the informed consent, female or male.
* Patients must have a Karnofsky performance status of 60 or more
* Patients must have limited systemic therapeutic options as per treating physician judgement. The number of previous lines of therapies is not limited.
* Patients with a tumor with a targetable oncogenic driver mutation should have already been treated with a targeted agent and options must have been exhausted.
* Patients must have a clinical indication for surgery for probable brain metastasis
* Patients will be considered eligible for the study only if the diagnosis of brain metastasis has been histologically confirmed on the sample obtained during the surgery performed after signing the informed consent form for the trial.
* Any type of primary cancer is allowed: breast cancer, lung cancer, melanoma, other cancers. Patients may have several primary cancers.
* Patients must have adequate bone marrow, renal and hepatic function documented at screening before surgery
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test
* Patients must have the ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
* Written informed consent for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention.

Exclusion Criteria:

* Patients with rapidly progressive systemic disease
* Patients with inability to undergo brain MRI evaluation.
* Patients with progressive parenchymal brain metastases with an indication for requiring whole brain radiotherapy after surgery. Focal brain radiotherapy after surgery is allowed.
* Judgement by the investigator that the patient is unlikely to comply with study procedures, restrictions and requirements.
* Intention to become pregnant during the course of the study.
* Female who are pregnant.
* Female who are breastfeeding and who do not agree to discontinue nursing prior to the first treatment initiated during the study.
* Sexually active males and females of childbearing potential who are not willing to use an effective contraceptive method during the study. Male participants who do not agree not to donate sperm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 8 months

SECONDARY OUTCOMES:
Response assessment | 8 months
  (A) in all patients: type of response; correlation of the type of response between CNS and extra-CNS compartments (B) in patients with measurable disease: type and duration of response; correlation of response rate between CNS and extra-CNS compartments.
Progression free survival | 8 months
Quality of life and neurological status 1 | 8 months
  EORTC-QLQ C30 scale
Quality of life and neurological status 2 | 8 months
  EORTC BN20 scale
Quality of life and neurological status 3 | 8 months
  NANO scale (Neurological Assessment in Neuro-Oncology)
Quality of life and neurological status 4 | 8 months
  Response assessement in Neuro-Oncology (RANO) seizure scale
Quality of life and neurological status 5 | 8 months
  Karnofsky performance status scale
Steroid use | 8 months
  Consumption of steroids during the study
Pharmacoscopy assessment 1 | 1 month
  rate of interpretable pharmacoscopy results, in the pharmacoscopy arm only
Pharmacoscopy assessment 2 | 1 month
  description of potential causes of failure of the pharmacoscopy analysis, in the pharmacoscopy arm only
Pharmacoscopy assessment 3 | 1 month
  rate of indication of pharmacoscopy guided-treatment, in the pharmacoscopy arm only
Pharmacoscopy assessment 4 | 1 month
  access to the preferred drug selected by the pharmacoscopy, in the pharmacoscopy arm only

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel
  - Cantonal Hospital St Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Weiss T, Buhler M, Mena J, Lottenbach Z, Wegmann R, Sun M, Bihl M, Augustynek B, Baumann SP, Goetze S, van Drogen A, Pedrioli PGA, Penton D, Festl Y, Buck A, Kirschenbaum D, Zeitlberger AM, Neidert MC, Vasella F, Rushing EJ, Wollscheid B, Hediger MA, Weller M, Snijder B. High-throughput identification of repurposable neuroactive drugs with potent anti-glioblastoma activity. Nat Med. 2024 Nov;30(11):3196-3208. doi: 10.1038/s41591-024-03224-y. Epub 2024 Sep 20. PMID 39304781
- [Background] Snijder B, Vladimer GI, Krall N, Miura K, Schmolke AS, Kornauth C, Lopez de la Fuente O, Choi HS, van der Kouwe E, Gultekin S, Kazianka L, Bigenzahn JW, Hoermann G, Prutsch N, Merkel O, Ringler A, Sabler M, Jeryczynski G, Mayerhoefer ME, Simonitsch-Klupp I, Ocko K, Felberbauer F, Mullauer L, Prager GW, Korkmaz B, Kenner L, Sperr WR, Kralovics R, Gisslinger H, Valent P, Kubicek S, Jager U, Staber PB, Superti-Furga G. Image-based ex-vivo drug screening for patients with aggressive haematological malignancies: interim results from a single-arm, open-label, pilot study. Lancet Haematol. 2017 Dec;4(12):e595-e606. doi: 10.1016/S2352-3026(17)30208-9. Epub 2017 Nov 15. PMID 29153976
- [Background] Kornauth C, Pemovska T, Vladimer GI, Bayer G, Bergmann M, Eder S, Eichner R, Erl M, Esterbauer H, Exner R, Felsleitner-Hauer V, Forte M, Gaiger A, Geissler K, Greinix HT, Gstottner W, Hacker M, Hartmann BL, Hauswirth AW, Heinemann T, Heintel D, Hoda MA, Hopfinger G, Jaeger U, Kazianka L, Kenner L, Kiesewetter B, Krall N, Krajnik G, Kubicek S, Le T, Lubowitzki S, Mayerhoefer ME, Menschel E, Merkel O, Miura K, Mullauer L, Neumeister P, Noesslinger T, Ocko K, Ohler L, Panny M, Pichler A, Porpaczy E, Prager GW, Raderer M, Ristl R, Ruckser R, Salamon J, Schiefer AI, Schmolke AS, Schwarzinger I, Selzer E, Sillaber C, Skrabs C, Sperr WR, Srndic I, Thalhammer R, Valent P, van der Kouwe E, Vanura K, Vogt S, Waldstein C, Wolf D, Zielinski CC, Zojer N, Simonitsch-Klupp I, Superti-Furga G, Snijder B, Staber PB. Functional Precision Medicine Provides Clinical Benefit in Advanced Aggressive Hematologic Cancers and Identifies Exceptional Responders. Cancer Discov. 2022 Feb;12(2):372-387. doi: 10.1158/2159-8290.CD-21-0538. Epub 2021 Oct 11. PMID 34635570